CLINICAL TRIAL: NCT00129194
Title: A Double-Blind, Placebo-Controlled, Dose Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of KP-1461 in HIV+ Adults Who Have Failed Two or More Highly Active Antiretroviral Regimens (HAART)
Brief Title: Study of KP-1461 for the Treatment of HIV Positive Patients Who Have Failed Multiple HAART Regimens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Koronis Pharmaceuticals. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KP-1461-102
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — KP 1461

INTERVENTIONS:
Drug: KP-1461

SUMMARY:
The primary purpose of the study is to assess the safety and pharmacokinetics of KP-1461 given every 12 hours for 14 days when administered to HIV+ patients who have failed multiple highly active antiretroviral therapy (HAART) regimens. Patients currently on HAART will be required to discontinue all HAART medications for up to 6 weeks after screening eligibility has been determined.

DETAILED DESCRIPTION:
KP-1461 is a carbamate prodrug of the active nucleoside, KP-1212. KP-1212 is incorporated into the proviral DNA. After multiple rounds of replication, KP-1212 increases the high inherent mutation rate of HIV beyond the threshold of viability, a process called "viral decay acceleration". KP-1212 is unique from conventional nucleoside reverse transcriptase inhibitors in that it inserts mutations randomly across the entire 10,000 nucleotide HIV genome and does not exert selective pressure by targeting a specific viral or cellular process, thus potentially avoiding drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* CD4 > 100 cells/mm3
* Viral load 2,500 - 200,000 copies/mL
* Exposure to at least 2 different HAART regimens containing NRTI(s), NNRTI(s), and 2 PI(s), excluding Ritonavir, for a minimum of 4 months or documented resistance to at least 3 of the 4 classes of approved antiretroviral drugs.
* Few, if any, effective treatment options available

Exclusion Criteria:

* HBsAb (hepatitis B) positive serology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Bach and Godofsky, Bradenton, Florida
  - University of Miami, Miami, Florida
  - Triple O Medical Services, West Palm Beach, Florida
  - Research Centers of Via Christi, Wichita, Kansas
  - Institute of Human Virology, University of Maryland, Baltimore, Maryland
  - Dybedal Center for Clinical Research, Kansas City University of Medicine and Biosciences, Kansas City, Missouri
  - St. Michael's Medical Center, Newark, New Jersey
  - AIDS Community Research Initiative of America, New York, New York
  - Greenville Hospital System, Greenville, South Carolina